CLINICAL TRIAL: NCT03642938
Title: The Dosing of Aerobic Exercise Therapy on Experimentally-induced Pain in Healthy Female Participants.
Brief Title: Exercise Dosing for Pain in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duquesne University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Benedict Kolber, Associate Professor, Duquesne University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-04-22; UL1TR001857 (NIH)
Record Dates: First submitted 2018-08-15; First posted 2018-08-22 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Pain
Keywords: Exercise; Dose; Analgesia
MeSH Terms: conditions — Pain; Motor Activity; Agnosia

STUDY DESIGN:
Intervention Model Description: Pseudo-randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose Exercise (Experimental): The Low Dose Exercise group will perform treadmill walking exercise, three times per week for one week.
  Interventions: Behavioral: Walking Exercise
- Moderate Dose Exercise (Experimental): The Moderate Dose Exercise group will perform treadmill walking exercise, five times per week for one week.
  Interventions: Behavioral: Walking Exercise
- High Dose Exercise (Experimental): The High Dose Exercise group will perform treadmill walking exercise, ten times per week for one week.
  Interventions: Behavioral: Walking Exercise
- Control (Sham Comparator): The Control group will perform quiet rest, three times per week for one week.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Walking Exercise — Exercise groups will perform moderate intensity treadmill walking at a speed of 3.5 mph at a 0% incline for 30 minutes.
  Arms: High Dose Exercise; Low Dose Exercise; Moderate Dose Exercise
Behavioral: Control — The Control group will perform 30 minutes of quiet rest.
  Arms: Control

SUMMARY:
In this study investigators will examine the effect of dose related to exercise therapy for pain in healthy adult humans. An acute pain model will be employed to study the effect of exercise dose on pain. Acute pain models are currently used to study pain (both acute and chronic) in human samples as there is currently no chronic pain model.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial with repeated measures. The effect of exercise dose on pain: subjects will be randomly assigned to one of four exercise groups: 1.) no exercise (control); 2.) low dose exercise (3x/week); 3.) moderate dose exercise (5x/week). 4.) high dose exercise (10x/week).

ELIGIBILITY:
Inclusion Criteria:

1. Between age 18-40
2. Normal BMI (18.5-25.0)
3. Heart Rate (HR) 60-100 bmp
4. BP less than or equal to 140/90

Exclusion Criteria:

1. Age <18 or >40 years
2. Cardiac, respiratory, neurological or musculoskeletal disease
3. Acute pain
4. Chronic pain condition
5. Diabetes
6. BMI ≥ 25.1 or ≤ 18.4
7. Regular participation in high intensity athletic/sporting activities
8. Sedentary
9. Anxiety or depression disorders
10. Tape allergy
11. Currently pregnant

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Szucs, PhD, Principal Investigator — Duquesne University; Amy L Phelps, PhD, Principal Investigator — Duquesne University; Matthew C Kostek, PhD, Principal Investigator — Duquesne University
Locations (1):
- Duquesne University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share. Raw data is available through the peer review publication.

REFERENCES:
- [Result] Polaski AM, Phelps AL, Szucs KA, Ramsey AM, Kostek MC, Kolber BJ. The dosing of aerobic exercise therapy on experimentally-induced pain in healthy female participants. Sci Rep. 2019 Oct 16;9(1):14842. doi: 10.1038/s41598-019-51247-0. PMID 31619738

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise | Control
Started | 10 | 10 | 10 | 11
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise | Control | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.7 (0.7) | 22.3 (3) | 20.6 (1.3) | 22.7 (3.7) | 21.58 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 10 | 10 | 40
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Intervention Effects on Mechanical Sensitivity Threshold
Description: Subjects' cutaneous mechanical sensitivity threshold will be examined using standard monofilaments that apply a force of 0.008g, 0.02g, 0.04g, 0.07g, 0.16g, 0.4g, 0.6g and 1.0g to the forearm and calf. Percent Baseline to 24 hrs post-intervention will then be calculated (100*Value at 24 hours/Value at Baseline). A filament of different weight is applied to the skin to look at the threshold of response.
Time Frame: baseline and 24 hrs-post final intervention session
Measure: Mean (Standard Error); unit: 100*Value at 24 hours/Value at Baseline
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise | Control
Number analyzed (Participants) | 10 | 10 | 10 | 10
100*Value at 24 hours/Value at Baseline
  Forearm Data | 125.6 (38) | 93.56 (36.03) | 63.04 (15.08) | 70.27 (23.15)
  Calf Data | 299 (138.9) | 396.7 (138.1) | 202.4 (65.09) | 287 (138.9)

2. Primary Outcome: Intervention Effects on Constant Heat Pain Intensity
Description: Subjects' constant heat pain intensity rating will be assessed using a (45 degree Celsius, 3cm x 5cm heating block applied to the forearm and calf for 3 seconds). Following the stimulus, subjects will rate the intensity of the pain associated with the stimulus using a visual analog scale numbered at 0 and 10, where "0" represents "no pain" and "10" represents "the worst pain imaginable" (0=minimum score, 10 maximum score). Percent baseline to 24 hrs post-intervention will then be calculated (100*Value at 24 hours/Value at Baseline).
Time Frame: baseline and 24 hrs-post final intervention session
Measure: Mean (Standard Error); unit: 100*Value at 24 hours/Value at Baseline
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise | Control
Number analyzed (Participants) | 10 | 10 | 10 | 10
100*Value at 24 hours/Value at Baseline
  Forearm | 88.79 (4.819) | 80.03 (21.37) | 80.16 (14.24) | 110.4 (55.20)
  Calf | 59.46 (9.12) | 114.3 (34.57) | 79.4 (22.68) | 136.3 (31.55)

3. Primary Outcome: Intervention Effects on Constant Heat Pain Unpleasantness
Description: Subjects' constant heat pain unpleasantness rating will be assessed using a (45 degree Celsius, 3cm x 5cm heating block applied to the forearm and calf for 3 seconds). Following the stimulus, subjects will rate the unpleasantness of the pain associated with the stimulus using a visual analog scale numbered at 0 and 10, where "0" represents "not unpleasant" and "10" represents "the most unpleasant sensation imaginable" (0=minimum score, 10 maximum score). Percent baseline to 24 hrs post-intervention will then be calculated (100*Value at 24 hours/Value at Baseline).
Time Frame: baseline and 24 hrs-post final intervention session
Measure: Mean (Standard Error); unit: 100*Value at 24 hours/Value at Baseline
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise | Control
Number analyzed (Participants) | 10 | 10 | 10 | 10
100*Value at 24 hours/Value at Baseline
  forearm | 110.1 (20.33) | 130.7 (48.24) | 110.6 (35.89) | 79.63 (39.68)
  calf | 65.94 (9.63) | 137.5 (33.49) | 83.20 (24.27) | 118.1 (39.50)

4. Primary Outcome: Intervention Effects on Radiant Heat Sensitivity
Description: Subjects' radiant heat sensitivity will be assessed using a temperature ramp from 30 degrees Celsius to 50 degrees Celsius over 60 seconds with participant defined cutoff in temperature (degrees Celsius) reading at their "sensitivity threshold" to the thermal stimulus (IITC Thermal Stimulus Apparatus with custom heated glass). This will be assessed on the forearm and calf. Percent baseline to 24 hrs post-intervention will then be calculated (100*Value at 24 hours/Value at Baseline).
Time Frame: baseline and 24 hrs-post final intervention session
Measure: Mean (Standard Error); unit: 100*Value at 24 hours/Value at Baseline
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise | Control
Number analyzed (Participants) | 10 | 10 | 10 | 10
100*Value at 24 hours/Value at Baseline
  forearm | 99.08 (1.4) | 101.2 (2.4) | 99.8 (1.46) | 100.8 (1.4)
  calf | 100.1 (2.68) | 101.5 (1.51) | 102.8 (3.10) | 102 (1.50)

5. Primary Outcome: Intervention Effects on Radiant Heat Pain
Description: Subjects' radiant heat pain threshold will be assessed using a temperature ramp from 30 degrees Celsius to 50 degrees Celsius over 20 seconds with participant defined cutoff in temperature (degrees Celsius) reading at their "pain threshold" to the thermal stimulus (IITC Thermal Stimulus Apparatus with custom heated glass). This will be assessed on the forearm and calf. Percent baseline to 24 hrs post-intervention will then be calculated (100*Value at 24 hours/Value at Baseline).
Time Frame: baseline and 24 hrs-post final intervention session
Measure: Mean (Standard Error); unit: 100*Value at 24 hours/Value at Baseline
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise | Control
Number analyzed (Participants) | 10 | 10 | 10 | 10
100*Value at 24 hours/Value at Baseline
  forearm | 98.65 (1.81) | 96.83 (3.14) | 97.10 (2.42) | 99.2 (2.60)
  calf | 100.6 (2.4) | 99.59 (1.7) | 104.5 (2.66) | 101.9 (1.999)

6. Primary Outcome: Intervention Effects on Pressure Pain Threshold
Description: Subjects' pressure pain threshold will be assessed using a pressure algometer (Wagner Instruments; 1cm round probe applied at constant ramping pressure until participant defined cutoff in kg at "pain threshold"). This will be assessed on the forearm and calf. Percent baseline to 24 hrs post-intervention will then be calculated (100*Value at 24 hours/Value at Baseline).
Time Frame: baseline and 24 hrs-post final intervention session
Measure: Mean (Standard Error); unit: 100*Value at 24 hours/Value at Baseline
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise | Control
Number analyzed (Participants) | 10 | 10 | 10 | 10
100*Value at 24 hours/Value at Baseline
  forearm | 135.5 (9.78) | 143.3 (14.01) | 150.1 (21.57) | 111 (9.01)
  calf | 122.6 (8.66) | 134.7 (10.02) | 130.8 (15.54) | 124.5 (12.65)

7. Primary Outcome: Intervention Effects on Constant Pressure Pain Intensity
Description: Subjects' constant pressure pain intensity rating will be assessed using a pressure algometer (Wagner Instruments; 1cm round probe applied for 2 seconds at participant defined threshold). Following the stimulus, subjects will rate the intensity of the pain associated with the stimulus using a visual analog scale numbered at 0 and 10, where "0" represents "no pain" and "10" represents "the worst pain imaginable" (0=minimum score, 10 maximum score). This will be assessed on the forearm and calf. Percent baseline to 24 hrs post-intervention will then be calculated (100*Value at 24 hours/Value at Baseline).
Time Frame: baseline and 24 hrs-post final intervention session
Measure: Mean (Standard Error); unit: 100*Value at 24 hours/Value at Baseline
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise | Control
Number analyzed (Participants) | 10 | 10 | 10 | 10
100*Value at 24 hours/Value at Baseline
  forearm | 93.3 (17.15) | 49.6 (6.87) | 67.26 (25.76) | 157.6 (20.83)
  calf | 89.6 (10.88) | 85.37 (33.67) | 74.30 (16.17) | 84.14 (11.23)

8. Primary Outcome: Intervention Effects on Constant Pressure Pain Unpleasantness
Description: Subjects' constant pressure pain unpleasantness rating will be assessed using a pressure algometer (Wagner Instruments; 1cm round probe applied for 2 seconds at participant defined threshold). Following the stimulus, subjects will rate the unpleasantness of the pain associated with the stimulus using a visual analog scale numbered at 0 and 10, where "0" represents "not unpleasant" and "10" represents "the most unpleasant sensation imaginable" (0=minimum score, 10 maximum score).This will be assessed on the forearm and calf. Percent change from baseline to 24 hrs post-intervention will then be calculated (100*Value at 24 hours/Value at Baseline).
Time Frame: baseline and 24 hrs-post final intervention session
Measure: Mean (Standard Error); unit: 100*Value at 24 hours/Value at Baseline
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise | Control
Number analyzed (Participants) | 10 | 10 | 10 | 10
100*Value at 24 hours/Value at Baseline
  forearm | 92.61 (17.34) | 46.62 (9.40) | 46.58 (14.6) | 127.9 (19.25)
  calf | 80.51 (9.95) | 76.56 (27.48) | 95.01 (36.24) | 114.7 (35.59)

9. Secondary Outcome: Heart Rate
Description: Heart rate will be measured before and after each exercise session. Percent pre-exercise session in heart rate (bpm) from start to end of exercise session will be calculated (100*Value at end trial/Value at start of trial).
Time Frame: days 1, 3, & 5 at start and end of each exercise session
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise
Number analyzed (Participants) | 10 | 10 | 10
Percent
  Day 1 | 124.12 (4.2) | 115.87 (7.15) | 112.349 (1.747)
  Day 3 | 121.443 (3.218) | 118.8 (5.7) | 110.16 (2.122)
  Day 5 | 113.440 (5.272) | 112.226 (4.632) | 109.221 (3.435)

10. Secondary Outcome: Borg Rate of Perceived Exertion (RPE)
Description: Subjects will indicate rate of perceived exertion before and after each exercise session. Percent of pre-exercise RPE from start to end of exercise session will be calculated (100* end of trial / start of trial).
Time Frame: days 1, 3, & 5 at start and end of each exercise session
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise
Number analyzed (Participants) | 10 | 10 | 10
Percent
  Day 1 | 144 (5.4) | 159.4 (8.1) | 152.45 (12.17)
  Day 3 | 147.2 (6.8) | 156.3 (7.12) | 161.3 (6.16)
  Day 5 | 154.6 (9.12) | 155.71 (7.11) | 157.98 (7.98)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during trial period only (1 week)
Description: Adverse events will be reported to IRB (Institutional Review Board).
Arm/Group | Low Dose Exercise | Moderate Dose Exercise | High Dose Exercise | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT03642938/Prot_002.pdf
  • Statistical Analysis Plan (2016-06-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT03642938/SAP_003.pdf